CLINICAL TRIAL: NCT03216161
Title: Sub-study for the Validation and Calibration of Data Regarding Physical Activity, Anthropometry and Diet
Status: Completed | Type: Observational
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Heiner Boeing, Head of the Department of Epidemiology, German Institute of Human Nutrition
Other Study IDs: 01ER0808
Record Dates: First submitted 2017-06-23; First posted 2017-07-13 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was an update and amplification of exposure measurements of the EPIC-Potsdam Study, which started in 1994-1998.

DETAILED DESCRIPTION:
The sub-study was conducted in the German Institute of Human Nutrition according to an approved study protocol.

The study program included comprehensive surveys on diet and lifestyle (smoking, physical activity, and anthropometry). The aim was to achieve repeated measurements in a sub-cohort of about 600 people to validate (measurement error correction) and calibrate (adjustment of insufficient data collected to the actual data location) existing baseline data in the entire cohort (EPIC-Potsdam cohort).

To this end, within age groups and by gender, active EPIC participants were then randomly selected in the years 2009 to 2012 from the cohort, contacted and invited to re-visit the respective study center. 816 subjects were acquired for re-examination, participation rate was 56.4%.

Each participant gave informed consent. The study protocol has been approved by the Ethics Committee of the Medical Association of the State of Brandenburg, Cottbus, on 18/12/2009.

The information in this section are study hypothesis and contains no results or conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the EPIC study who meet the following three conditions were eligible for invitation to the re-examination:

  1. actively participating in the EPIC-Potsdam follow-up
  2. current address in Brandenburg or Berlin
  3. phone number known

Exclusion Criteria:

* Not meeting the above stated criteria

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Potential participants were drawn from the cohort study population in the EPIC-Potsdam Study based on a gender- and age-stratified random sample and invited successively.
  First stage: gender (male / female, 300 each) Second stage: the age at recruitment to EPIC Potsdam (35-44y/ 45-54y/ 55-64; 100 each)
Study Population: Participants of the EPIC-Potsdam cohort study were 35-64 years old at recruitment (1994-1998). For this study (re-examination 2010-2012), participants were 47-81 years old (mean age 65.5, were largely sedentary and with a mean BMI of 27.5 kg/m2). Participants were living in the state of Brandenburg or in Berlin, Germany.
  The information in this section are study hypothesis and contains no results or conclusions.
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improved and more detailed assessment of food intake | 4-24 months
  Repeated 24 hour dietary recalls. Every participant provided up to three (mean = 2.99) 24 hour dietary recalls at baseline (cross-sectional analysis). The recalls were performed by trained interviewers using EPIC-Soft program and were collected within a period of 4-24 months (mean = 7). The first recall took place in person during the participants' first visit to the study center. The following two recalls took place on random days over the telephone. Food consumption was recorded in 11 eating occasions (before breakfast, breakfast, after breakfast, during morning, lunch, after lunch, during the afternoon, before dinner, dinner, after dinner, during evening) and was recorded for each food in grams per eating occasion.

SECONDARY OUTCOMES:
Body weight | Appointment at the study center at beginning of study
  In kilograms. For the purpose of achieving improved and more detailed assessment of anthropometric measeures
Skinfold thickness | Appointment at the study center at beginning of study
  In millimeters. For the purpose of achieving improved and more detailed assessment of anthropometric measeures
Magnetic resonance imaging (MRT) | Within 4 weeks after first visit to the study center
  The measurements were performed with a 1.5T MRT scanner ("Magnetom Avanto", Siemens, Erlangen, Germany) and the Vibe Dixon sequence. The Vibe-Dixon sequence is a special MRT protocol fornbody fat analysis which separates the fat from tissue water. Fat tissue is displayed brightly, while the remaining tissue appears dark.
Other anthropometric measures | Appointment at the study center at beginning of study
  Height, circumference of hip and waist, depth and width of chest (all in centimeters). For the purpose of achieving improved and more detailed assessment of anthropometric measeures
Physical activity level (PAL) | 1 week
  A heart rate monitor and integrated accelerometer ("Actiheart" CamNtech, Cambridge, UK) was work for a week of everyday life. The Actiheart software calculated physical activity based on the individual calibration models in the form of "Physical Activity Levels", which is the ratio of the total energy expenditure for resting enery expenditure.
Physical activity questionnaire | 12 months (retrospective questionnaire)
  Participants also filled in a questionnaire on physical activity (physical activity during the past 12 months and activities in the last 4 weeks).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neamat-Allah J, Wald D, Husing A, Teucher B, Wendt A, Delorme S, Dinkel J, Vigl M, Bergmann MM, Feller S, Hierholzer J, Boeing H, Kaaks R. Validation of anthropometric indices of adiposity against whole-body magnetic resonance imaging--a study within the German European Prospective Investigation into Cancer and Nutrition (EPIC) cohorts. PLoS One. 2014 Mar 13;9(3):e91586. doi: 10.1371/journal.pone.0091586. eCollection 2014. PMID 24626110
- [Background] Wientzek A, Vigl M, Steindorf K, Bruhmann B, Bergmann MM, Harttig U, Katzke V, Kaaks R, Boeing H. The improved physical activity index for measuring physical activity in EPIC Germany. PLoS One. 2014 Mar 18;9(3):e92005. doi: 10.1371/journal.pone.0092005. eCollection 2014. PMID 24642812